CLINICAL TRIAL: NCT05041595
Title: Collection of Whole Blood to be Used to Provide the Safety and Effectivenss of a Lyme Disease Diagnostic Assay to Support the Proposed Intended Use Statement and Product Labeling Claims.
Brief Title: Lyme Disease Diagnostic Assay - Collection of Whole Blood
Status: Enrolling by invitation | Type: Observational
Sponsor: DiaSorin Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROT.648.00024.A
Record Dates: First submitted 2021-08-26; First posted 2021-09-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Lyme Disease; Healthy
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Sick Cohort: Borreliosis Subjects - All comers expressing signs and symtoms consistent with suspicion of acute Borreliosis and under medical examination for Lyme disease Borreliosis subjects with an Erythema Migrans Rash (subgroup)
  Interventions: Diagnostic Test: Lyme diagnostic assay
- Apparently Healthy: Apparently healthy subjects living in an area non-endemic for Lyme disease Apparently healthy subjects living in an area endemic for Lyme disease
  Interventions: Diagnostic Test: Lyme diagnostic assay

INTERVENTIONS:
Diagnostic Test: Lyme diagnostic assay — Serological and immunoresponse assay

SUMMARY:
The primary objective is to obtain whole blood from subjects with signs and/or symptoms of early Borrelisois. Whole blood will also be obtained from subjects with suspicion of acute Borreliosis and under medical examination for Lyme disease.

In addition, whole blood will be obtained from apparently healthy subjects residing in areas endemic to Lyme disease and may also inlclude apparently healthy subjects residing in areas non-endemic to Lyme disease.

DETAILED DESCRIPTION:
Whole blood will be collected, and processed. Some blood will be transferred to additional tubes for further processing and aliquotting. Serum and plasma will be harvested and tested, at a later date, in a clinical performance study with approved and/or commercially available devices as well as an investigational Lyme assay. This study will be coordinated by the Sponsor.

ELIGIBILITY:
Subjects with under evaluation of Lyme Disease

Inclusion Criteria:

Signs and symptoms of acute Lyme disease which include at least one of the following:

* Recent onset of fatigue
* Skin rash
* Fever
* Muscle aches
* Neck pain
* Joint pain or lymphadenopathy

Subgroup Borreliosis Subjects- restricted signs and symptoms of acute Lyme including EM Rash

* Under physician or medical evaluation for acute on-set of Lyme Disease presenting with EM Rash
* Detailed description of the EM rash (e.g. Itchy, painful, hot, vesicular, raised) with consent for photographic documentation is required including additional picture with ruler placing to confirming size.
* EM rash with the following attributes:

  * Size > 5 cm in diameter
  * Appeared 3-30 days after bite or suspected bite
* Specify Location (e.g. underarm or back of knee)
* Subjects with confirmed early localized or disseminated Lyme Borreliosis manifestation
* Signs and symptoms (e.g. Fever, Chills/Sweats, Headache, Fatigue/Tiredness, Myalgia/Sore muscles)
* The EM rash has been present <42 days
* Clinical diagnosis of Lyme disease is suspected by the practitioner
* Ability to provide the minimum sample volume required

Exclusion Criteria:

* Subjects unable to provide informed consent.
* Subjects without clinical information and/or not meeting inclusion criteria.
* Subjects having started antibiotic treatment > 5 days before inclusion.

Healthy Subjects

Inclusion Criteria:

* Apparently healthy subjects with no present fever, chills, headache, fatigue, muscle and joint aches, and swollen lymph nodes, e.g. flu-like symptoms.
* Ability to provide the minimum sample volume required.

Exclusion Criteria:

- ● Subjects unable to provide informed consent

* Subjects without clinical information and/or not meeting inclusion criteria
* Subjects with a recent diagnosis of Lyme disease, Anaplasmosis, Babesiosis, or history of known embedded tick bite which may have required 'manual extraction' NOTE: a tick just found on the subject or presence of a crawling tick is not considered a 'tick bite')
* Subjects currently on antibiotic treatment.
* Uncontrolled HIV-infection, if known. This is defined as an HIV-1 viral load >40 copies/mL and/or CD4+ count <500 x 106 cells/liter in the past 12 months.
* Active syphilis or leptospirosis, if known
* Active infection with Epstein Barr Virus (mononucleosis), if known
* Active infection with Cytomegalovirus (CMV), if known
* Subjects with autoimmune diseases, either confirmed rheumatoid arthritis and/or other autoimmune disorders diagnosed according to the leading guidelines
* Current immunomodulation mediation including >7.5 mg prednisone daily, methotrexate, and/or biologicals. Medications such as hydroxychloroquine, sulfasalazine or NSAIDs are acceptable.
* Immunodeficiency, hematologic malignancies in the medical history
* Chemotherapy during the past year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with suspected Borreliosis including subjects with EM rash and subjects without EM rash but with signs and symptoms consistent with suspicion of acute Borreliosis and under medical examination for Lyme disease.
  Healthy subjects living in endemic Lyme disease area and healthy subjects living in a non-endemic Lyme disease area.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance - Sensitivity | Through study completion, an average of 1 year
  Diagnostic Sensitivity

SECONDARY OUTCOMES:
Clinical Performance - Specificity | Through study completion, an average of 1 year
  Diagnostic Specificity

CONTACTS AND LOCATIONS:
Locations (1):
- DiaSorin Inc., Stillwater, Minnesota, United States